CLINICAL TRIAL: NCT01186822
Title: A Six Month Randomized Controlled Clinical Trial of Lung Flute in Patients With Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaas J Smit PhD (Industry)
Responsible Party: Sponsor-Investigator, Nicolaas J Smit PhD, Dr. S. Sethi, Medical Acoustics LLC
Organization: Medical Acoustics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LF6mo
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung Flute for BHT (Experimental): The Lung Flute arm participants were instructed to blow twice in to the Lung Flute device vigorously enough to make the reed oscillate, followed by 5 normal breaths. This was repeated 10 times, followed by 3 huff coughs to complete 1 cycle. Two such cycles were recommended twice a day. One of these cycles was performed under supervision of the study personnel at the time of enrollment and at each subsequent study visit. Baseline COPD medication regimen was continued in all participants, although the primary physicians of the participants could make medically necessary changes. Chest physical therapy, additional breathing exercises and formal pulmonary rehabilitation programs were not prescribed to any of the participants during the study.
  Interventions: Device: Lung Flute
- No intervenstion (No Intervention): No intervention. Same population.

INTERVENTIONS:
Device: Lung Flute — Used twice daily
  Arms: Lung Flute for BHT

SUMMARY:
This is a 26 week randomized controlled study. The study consists of, in order, an enrollment visit, followed by clinic visits at 2 weeks, 14 weeks and at 26 weeks. There will also be telephonic assessments at 8 weeks and 20 weeks. Clinic visits will involve comprehensive assessments of the patients lung condition, including post-bronchodilator spirometry, Shuttle walk distance, BODE index, health status (SGRQ) and symptoms (CCQ). Sputum and serum samples will also be collected at these visits for microbiological and inflammation analysis. Sputum will be obtained with the Lung Flute as an induction device and Pulse Oximetry will be assessed prior to and after use of the Lung Flute. Clinic and telephonic visits will collect information regarding compliance with the use of the Lung Flute, adverse events and exacerbation history.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between and including the ages of 30 and 80 years. Females of childbearing potential may be included provided they are not pregnant or are not nursing.
2. Subjects with a diagnosis of moderate to very severe chronic obstructive pulmonary disease as defined by the Global Initiative for COPD (GOLD, 2008 update) and who meet the following criteria for stage ll - IV disease:

   a) Subjects must have a post-bronchodilator FEV1/FEV ratio <70% and FEV1 of <80% of the predicted value for age, height, and sex using the NHANES III standards (Hankinson, 1999).
3. Subjects must have a smoking history of at least 10 pack-years.
4. Subjects must have stable disease for at least 1 month prior to enrollment with no changes in the maintenance treatment for COPD in this period.

   -

Exclusion Criteria:

1. History of an exacerbation or other significant disease instability during the month preceding enrollment.
2. A primary diagnosis of asthma or bronchiectasis.
3. Inability to vibrate the reed of the Lung Flute® consistently because of severely expiratory flow rate.
4. Subject with any evidence of significant concomitant clinical disease that, in the opinion of the investigator, could interfere with the conduct of the study or safety of the subject.
5. Pregnant or nursing females or females intending to become pregnant during the course of the study.
6. Use of any investigational drug within one month or 6 half-lives (which-ever is greater) of the enrollment visit.
7. Inability to comprehend or willingness to follow the study requirements including attendance at out-patient clinic visit and participation in testing as called for by the protocol.
8. Patients currently using the Lung Flute. -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in COPD symptoms assessed by the CCQ questionnaire between the intervention and control group. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sethi, MD, Principal Investigator — VA WNY Healthcare System
Locations (1):
- VA WNY Healthcare System, Buffalo, New York, United States

REFERENCES:
- [Derived] Sethi S, Yin J, Anderson PK. Lung flute improves symptoms and health status in COPD with chronic bronchitis: A 26 week randomized controlled trial. Clin Transl Med. 2014 Sep 23;3:29. doi: 10.1186/s40169-014-0029-y. eCollection 2014. PMID 25625006